CLINICAL TRIAL: NCT00043654
Title: Antiglucocorticoid Therapy in Bipolar Depression With Mifepristone (RU486)
Brief Title: Clinical Trial of Mifepristone for Bipolar Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 020251; 02-M-0251
Record Dates: First submitted 2002-08-09; First posted 2002-08-12 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-06-25

CONDITIONS: Bipolar Disorder
Keywords: Antidepressant; Manic-Depressive Disorder; Cortisol; Neuroendocrine; Cognition; Bipolar; Bipolar Disorder; BPD; HV
MeSH Terms: conditions — Bipolar Disorder | interventions — Mifepristone

INTERVENTIONS:
Drug: Mifepristone

SUMMARY:
Bipolar Depression is a severe illness with high rates of psychiatric comorbidity and increased mortality related to suicide and medical illness. Hypothalamic pituitary axis (HPA) hyperactivity are found in bipolar disorder related to depression and mixed states. Patients with bipolar disorder also have cognitive difficulties and endocrine disturbances may contribute to such dysfunction. Antiglucorticoid therapies are novel treatments of mood disorder. Preliminary data in psychotic depression suggesting that mifepristone (RU-486), a glucocorticoid receptor antagonist, has antidepressant and salutary cognitive effects in a matter of days. In this study we examine the effects of mifepristone in severe bipolar depression in a parallel, double blind placebo controlled experiment. Bipolar subjects maintained on either lithium or valproate, after washout or prior antidepressants have a detailed neuroendocrine assessment. Patients approximately or almost 75 will receive eight days of mifepristone versus placebo after which patients are blindly crossed over to the opposite arm. Patients and a group of matched controls approximately or almost 35 will be compared with neuroendocrine, cognitive, and neurophysiologic testing to fully characterize their phenotype and explore biomarkers of response. It is hypothesized that stigmata of HPA axis hyperactivity and cognitive impairment will be predictive of response to antiglucocorticoid therapy with mifepristone.

DETAILED DESCRIPTION:
Bipolar Depression is a severe illness with high rates of psychiatric comorbidity and increased mortality related to suicide and medical illness. Hypothalamic pituitary axis (HPA) hyperactivity are found in bipolar disorder related to depression and mixed states. Patients with bipolar disorder also have cognitive difficulties and endocrine disturbances may contribute to such dysfunction. Antiglucorticoid therapies are novel treatments of mood disorder. Preliminary data in psychotic depression suggesting that mifepristone (RU-486), a glucocorticoid receptor antagonist, has antidepressant and salutary cognitive effects in a matter of days. In this study we examine the effects of mifepristone in severe bipolar depression in a parallel, double blind placebo controlled experiment. Bipolar subjects maintained on either lithium or valproate, after washout or prior antidepressants have a detailed neuroendocrine assessment. Patients approximately or almost 75 will receive eight days of mifepristone versus placebo after which patients are blindly crossed over to the opposite arm. Patients and a group of matched controls approximately or almost 35 will be compared with neuroendocrine, cognitive, and neurophysiologic testing to fully characterize their phenotype and explore biomarkers of response. It is hypothesized that stigmata of HPA axis hyperactivity and cognitive impairment will be predictive of response to antiglucocorticoid therapy with mifepristone.

ELIGIBILITY:
* HEALTHY VOLUNTEERS ARE CURRENTLY NOT BEING RECRUITED FOR THIS STUDY.

INCLUSION CRITERIA FOR BIPOLAR PATIENTS:

Patients must meet the following inclusion criteria in order to participate in the study:

1. Male or female inpatients in need of treatment for severe bipolar depression.
2. 18-75 years of age.
3. Women of childbearing potential must be using an adequate form of contraception as defined by one of the following: 1) a barrier method and 2) oral contraceptives plus a barrier method (women who are on an OCP will be kept on it others must agree to use only a barrier method).
4. DSM-IV diagnosis of bipolar depression I/II, severe, with or without psychotic features.
5. A current major depressive episode of at least 6 weeks' duration.
6. Score of greater than or equal to 18 on the first 17-item HAM-D at the prestudy visit and at the first baseline phase visit.
7. Score of 15 or greater on the HAM-D (17) at the end of the baseline period(s) (i.e., at randomization no more than 20% less than entry enrollment criteria).
8. Score of greater than or equal to 4 on the CGI-BP scale at the prestudy and first visit and end of baseline phase.
9. Judged to be in good physical health on the basis of medical history, physical examination, and laboratory screening.
10. Able to understand procedures and agree to participate in the study by giving written informed consent.
11. On lithium and/or valproate for at least 4 weeks (2 levels, 1 wk apart)
12. However patients not on a mood stabilizer can have this started as an outpatient or inpatient for 4 weeks as discussed above.
13. Able to come off of prior drugs and PRN zolpidem and lorazepam by start of baseline.

EXCLUSION CRITERIA FOR BIPOLAR PATIENTS:

Patients will be excluded from the study if they meet any of the following criteria:

1. Women who are pregnant, intending to become pregnant in the next month or breast-feeding.
2. Treatment with any of the following therapies within the specified interval prior to baseline: Fluoxetine - 4 weeks; Investigational compounds 4 weeks; MAOIs 1 week; Other antidepressants 1 week.
3. Contraindication or history of hypersensitivity to mifepristone as well as cortisol, and CRH.
4. Clinically significant organ system disease where mifepristone would be contraindicated or interfere with medical treatment.
5. Have evidence of any disorder that represents a contraindication to the use of mifepristone (such as adrenal disease or a condition requiring chronic corticosteroid administration).
6. History of Addison's Disease, Cushing's Disease, insulin dependent diabetes, or other uncompensated endocrine conditions.
7. Evidence of infection, severe liver, respiratory, or renal disease.
8. Have clinically significant cardiovascular disease, e.g., angina, valve disease, arrhythmia, cardiac failure.
9. Anemia (hemoglobin less than 10 g/dL or hematocrit less than 30%)
10. Have a known clotting defect or are receiving anticoagulants.
11. Rapid cycling in the last year (defined as greater than 6 episodes).
12. History of porphyrias.
13. Clinically significant abnormalities in physical exam, ECG, or laboratory assessments.
14. History of any disease which, in the investigator's opinion may confound the results of the study or pose an additional risk, including but not limited to, history of organic mental disorder, seizures, or mental retardation.
15. Substance dependence that is not in sustained full remission (DSM-IV definition)
16. Other principal psychiatric diagnosis judged by the investigator to dominate the clinical presentation. In particular, patients with depressive symptoms more than 2 years in duration should be carefully evaluated to determine whether another psychiatric diagnosis exists which could interfere with efficacy and safety measurements.
17. History of nonresponse to greater than four trials of antidepressants for the current episode (not including mood stabilizers) will exclude subjects.

INCLUSION CRITERIA FOR NORMAL CONTROLS:

1. SCID-NP- no psychiatric diagnosis lifetime.
2. Ages 18-75.
3. Medically and psychiatrically healthy by history and no disallowed medications for 2 weeks, and agrees to no alcohol use for 1 week baseline period of study.
4. No history of mood or anxiety disorder in first-degree relatives.
5. Women of childbearing potential must be using adequate form of contraception as defined by one of the following: 1) a barrier method and 2) oral contraceptives plus a barrier method.

EXCLUSION CRITERIA FOR NORMAL CONTROLS:

1. Known hypersensitivity to CRH, hydrocortisone, metyrapone, or mifepristone.
2. Women who are pregnant or breast-feeding.
3. Clinically significant organ system disease where mifepristone would be contraindicated or interfere with medical treatment.
4. History of prophyrias.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110
Dates: Start 2002-08-07; Study Completion 2007-06-25

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Sapolsky RM. Stress, Glucocorticoids, and Damage to the Nervous System: The Current State of Confusion. Stress. 1996 Jul;1(1):1-19. doi: 10.3109/10253899609001092. PMID 9807058